CLINICAL TRIAL: NCT00206986
Title: Will Decreased Noradrenergic Activity Normalize Information Processing in Patients With Schizophrenia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birte Glenthoj (Other)
Collaborators: University of Copenhagen (Other); Lundbeck Foundation (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 363037-2; KF 11-261729
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Information processing; PPI; P50 gating; P300; mismatch negativity; clonidine
MeSH Terms: conditions — Schizophrenia | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: clonidine
- 2 (Experimental)
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — Either placebo or 25 ug, 50 uG 75 ug or 150 ug of clonidine will be added to the current medication of patients with schizophrenia, who are stable on their current medication
  Other Names: Catapressan
  Arms: 1
Drug: clonidine — 0.15 mg of clonidine will be administered to 20 healthy male volunteers
  Other Names: Catapressan
  Arms: 2

SUMMARY:
The investigators want to try to improve information processing in schizophrenic patients via pharmacological intervention. The hypothesis is that decreased noradrenergic activity will normalize information processing (PPI, P50 gating, P300, and mismatch negativity) in patients with schizophrenia.

DETAILED DESCRIPTION:
A number of reports in literature provide evidence for, among others, an increased central noradrenergic activity in schizophrenia. In addition to this increased noradrenergic activity, patients with schizophrenia often show reduced filtering of sensory information, which is reflected in reduced P50 suppression and reduced prepulse inhibition of the startle reflex (PPI). In two separate initial studies in our laboratory, we found reduced sensory gating following administration of imipramine (a combined noradrenergic and serotonergic agonist) and desipramine (a highly specific noradrenergic agonist) to healthy volunteers. This provides evidence for a direct causal relation between the increased noradrenergic activity and the disturbed gating of sensory information, as both commonly found in patients with schizophrenia. Therefore, in a follow-up study, the effects of a noradrenergic antagonist will be investigated on the sensory gating of patients with schizophrenia. To further extend the data of our initial studies, the patients will additionally be tested for two psychophysiological parameters of attention that are usually found to be disturbed in patients with schizophrenia, i.e. mismatch negativity and selective attention. The design will conform to a double blind, placebo controlled experiment, in which either four doses (0.25 ug, 50 ug, 75 ug or 150 ug)of clonidine or placebo will be added to the current medical treatment of 20 male patients with schizophrenia on five occasions, separated by at least a week, after which they are tested in the Copenhagen Psychophysiological Test Battery (CPTB).In order to test the effects of clonidine in healthy volunteers, 20 healthy males will receive a fixed dose of 0.15 mg clonidine or placebo on two separate occasions separated by at least a week, after which they will be tested in the CPTB as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Male subjects
  * Meeting the DSM-IV diagnosis of schizophrenia
* Controls:

  * Male subjects
  * Good Physical and Mental Health meeting criteria "never mentally ill", which will be evaluated with a medical history checklist
  * Non smokers

Exclusion Criteria:

* Patients:

  * A P50 suppression or PPI score falling within a range of 10 percent above or below the mean score of the healthy control group
* Controls:

  * Current use of any medication
  * Any subject who has received any investigational medication within 30 days prior to the start of this study
  * History of neurologic illness
  * History of psychiatric illness in first-degree relatives, evaluated with DSM-IV criteria
  * History of alcohol and drug abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The following psychophysiological measures: | prospective
Prepulse Inhibition og the Startle Response (PPI) | Once, 3.5 hrs after intake of capsule
P50 suppression | Once, 3.5 hrs after intake of capsule
P300 Event Related Potential | Once, 3.5 hrs after intake of capsule
Mismatch negativity | Once, 3.5 hrs after intake of capsule
PANSS | 5 times hourly after intake of capsule

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc., Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychaitric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Copenhagen NV, Denmark

REFERENCES:
- See also: Center for Neuropsychiatric Schizophrenia Research (CNSR) — http://www.cnsr.dk